CLINICAL TRIAL: NCT00923442
Title: Hematologic Malignancy Biology Study
Brief Title: Biology Studies of Hematologic Cancers
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040102; 04-C-0102; NCT00900393 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-18

CONDITIONS: Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome (MDS); Non-Hodgkins Lymphoma; Acute Myelogenous Leukemia; Hodgkins Lymphoma
Keywords: Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia; Pediatric Blood Disorders; Hodgkins and non-Hodgkins lymphoma; MDS; Natural History
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: patients (from >/= 1 to 75 years old) diagnosed with any hematologic malignancy or pre-malignant condition

SUMMARY:
This study will collect tumor samples from people with cancers of the blood, bone marrow, or lymph glands for laboratory study of the biology of these conditions. Such studies contribute to a better understanding of cancer biology and to the development of new treatments. Planned studies include:

* Examination of individual cancer cells and to search for differences compared to other types of cancer and normal cells
* Examination of the chromosomes and genes in cancer cells and to search for differences compared to other types of cancer and normal cells
* Development of sensitive methods to detect small amounts of cancer that remain after treatment
* Search for new cancer proteins that might serve as targets for treatment
* Investigation of methods to develop cancer vaccines.

Patients from >= 1 to 75 years of age with acute lymphocytic leukemia, acute myelogenous leukemia, myelodysplastic syndrome, chronic myelogenous leukemia, juvenile myelomonocytic leukemia, non-Hodgkin's lymphoma, Hodgkin's disease, and other hematologic malignancies may be eligible for this study.

Blood or bone marrow samples will be collected when sampling is required for the patient's medical care. Cells from some individuals will be grown in test tubes, establishing cell lines or in animals, establishing xenograft models. (A xenograft is transplantation of cells of one species to another species.)

DETAILED DESCRIPTION:
Background:

Laboratory-based investigations have contributed to an improved understanding of pathophysiology and to the development of new therapies for hematologic malignancies.

The aim of this protocol is to facilitate biologic study of leukemias, pre-malignant conditions, myelodysplastic syndromes, lymphomas, and other blood disorders.

This is a sample acquisition protocol for targeted study of hematologic malignancies by a collaborative network of NIH investigators from multiple Institutes/Centers.

Objective:

This biology protocol is designed to allow sample acquisition for use in the study of hematologic malignancies. A variety of laboratory investigations designed to support NIH translational trials, to apply new methodologies in the study of cellular, and molecular biology, to probe for new therapeutic targets; and to develop new treatment approaches will be performed.

Eligibility:

Diagnosis of any hematologic malignancy or pre-malignant conditions, including but not restricted to the following: Acute Lymphocytic Leukemia (ALL), Acute Myelogenous Leukemia (AML), Myelodysplastic Syndrome (MDS), Chronic Myelogenous Leukemia (CML), Juvenile Myelomonocytic Leukemia (JMML, J-CML), Non-Hodgkin s Lymphoma (NHL), Hodgkin s Disease

Tumor tissue that has been previously collected and is available for study or that can be collected with minimal additional risk to the subject during sampling required for routine patient care.

Patient age: >= 1 year

Design:

Biologic assays relevant to the investigation of hematologic malignancies will be performed in an exploratory fashion, some studies are developmental, i.e., assay design in support of current or planned CC clinical trials. Others are standard assays that will be applied in attempt to identify new targets or test new therapeutic approaches.

.

ELIGIBILITY:
* INCLUSION CRITERIA

Confirmed pathological diagnosis of any hematologic malignancy or pre-malignant blood disorder, including but not restricted to the following:

Acute Lymphocytic Leukemia (ALL)

Acute Myelogenous Leukemia (AML)

Myelodysplastic Syndrome (MDS)

Chronic Myelogenous Leukemia (CML)

Juvenile Myelomonocytic Leukemia (JMML, J-CML)

Non-Hodgkin's Lymphoma (NHL)

Hodgkin's Disease

Tumor tissue that has been previously collected and is available for study or that can be collected with minimal additional risk to the subject during sampling required for routine patient care.

Age: >= 1 years.

Prior therapy: no restrictions

Subject, parent/guardian, legally authorized representative (LAR), or durable power of attorney must be able to give informed consent and sign the informed consent document.

EXCLUSION CRITERIA

None

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tumor tissue of patients whose ages range from birth to 75 years old diagnosed with any hematologic malignancy or pre-malignant blood disorder
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2004-02-24 (Actual)

PRIMARY OUTCOMES:
Tissue acquisition for lab investigations | 1 Month
  The examination of biologic assays relevant to the investigation of hematologic malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-C-0102.html